CLINICAL TRIAL: NCT07374640
Title: Virtual Reality and Biofeedback for Adolescents With Chronic Dizziness
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Jacob Brodsky, Director, Balance & Vestibular Program, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-P00041413
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Persistent Postural Perceptual Dizziness; Vestibular Migraine; Chronic Dizziness
Keywords: Persistent Postural-Perceptual Dizziness; Vestibular Migraine; Chronic Dizziness; Virtual Reality; Biofeedback

STUDY DESIGN:
Intervention Model Description: This is a pilot study evaluating the feasibility and effectiveness of VR as an addition to the standard-of-care treatments of BFB, SDERP, and CBT for treating chronic dizziness and PPPD in adolescents.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- VR in conjunction with BFB, SDERP, and CBT (Experimental): This group will undergo virtual reality exercises in conjunction with the standard-of-care biofeedback, systematic desensitization exposure response prevention, and cognitive behavioral therapy.
  Interventions: Device: Virtual Reality

INTERVENTIONS:
Device: Virtual Reality — Application of a virtual reality headset and experience in a virtual realty environment in addition to the standard-of-care biofeedback, systematic desensitization exposure response prevention, and cognitive behavioral therapy.
  Other Names: VR

SUMMARY:
Both persistent postural-perceptual dizziness (PPPD) and vestibular migraine (VM) are common diagnoses in patients presenting to physicians for evaluation of vestibular symptoms such as dizziness and vertigo. Although they are most often described in the adult population, they are also common in children and adolescents with dizziness. Chronic dizziness profoundly affects quality of life, often keeping children out of school and inhibiting their participation in the normal activities of childhood and adolescence. Overall, chronic dizziness is suspected to be due in large part to a "rewiring" of the brain that alters how cues related to balance and orientation are processed, with overreliance on visual inputs to maintain balance and equilibrium being a common development. Thus, chronic dizziness, especially that which is due to PPPD, is often caused by visual triggers.

A multi-modal approach is often taken to treat chronic dizziness, attempting to recalibrate this maladaptive "rewiring" and return the sensory system to normal function. Given the role that visual inputs play in developing and perpetuating chronic dizziness, habituation to visual stimuli should be a significant component to treatment. Treatments often include cognitive behavioral therapy (CBT), systematic desensitization exposure response prevention (SDERP), and biofeedback therapy (BFB). However, these visually provoked symptoms are often resistant to treatment. One reason for this may be that visual stimuli are difficult to replicate in the clinic or office. One way to address this gap in treatment is through virtual reality (VR) technology, which immerses patients in realistic visual environments.

VR has not been explicitly described in the treatment of PPPD or chronic dizziness, but it has been piloted, and shown to be effective, in the rehabilitation of peripheral vestibular dysfunction. This study aims to integrate VR into the current PPPD/chronic dizziness techniques of CBT, SDERP, and BFB. We will use a commercially available VR headset, which enables the use of VR in the office setting in a relatively low-cost form of VR technology. This study will evaluate the feasibility and effectiveness of VR in conjunction with CBT, SDERP, and BFB to investigate if VR technology enhances previously established effective treatments to reduce chronic dizziness and PPPD.

DETAILED DESCRIPTION:
Persistent postural-perceptual dizziness (PPPD) is a chronic vestibular disorder characterized by dizziness, unsteadiness, or non-spinning vertigo exacerbated by position changes, active or passive motion, and complex or moving visual stimuli. PPPD was defined in 2017 as an addition to the International Classification of Vestibular Disorders and will be included in the next iteration of the International Classification of Diseases by the World Health Organization (ICD-11). It is a common diagnosis in patients presenting to tertiary centers for evaluation of vestibular symptoms. Although PPPD is most often described in the adult population, it is also common in children and adolescents with dizziness.

Vestibular migraine is the most common cause of episodic dizziness in children and adults. It can sometimes cause chronic, daily dizziness symptoms and can sometimes also trigger concurrent PPPD, which also causes chronic, daily dizziness.

The symptoms of chronic dizziness profoundly affect quality of life, often keeping children out of school. Moreover, most patients are symptomatic for many months or even years before receiving a diagnosis and initiating treatment. As PPPD is not likely to resolve spontaneously or without treatment, effective early treatment is crucial to alleviating symptom burden. Chronic vestibular migraine is typically treated primarily with medications, which can cause side effects and are sometimes inadequate to achieve complete symptom control.

PPPD is typically precipitated by an event that causes dizziness, vertigo, or unsteadiness, such as an acute or episodic peripheral vestibular disorder, concussion, psychological distress, or adverse medication effect. Though an utterly definitive model is still being established, it is widely accepted that PPPD may develop following these inciting events through the development and perpetuation of maladaptive compensatory strategies, such as overreliance on visual inputs to maintain equilibrium and balance, and heightened anxiety or body vigilance during self-motion or motion-rich environments. These responses to dizziness or unsteadiness are typically transient but become persistent and maladaptive in PPPD, leading to a "rewiring" of the brain that alters how cues related to balance and orientation are processed.

A multi-modal approach to chronic dizziness treatment is often taken to recalibrate maladaptive compensatory strategies and return the sensory system to normal function. One component of treatment includes cognitive behavioral therapy (CBT). The overall goals of CBT include reducing behaviors, thoughts, feelings, and symptoms that perpetuate chronic dizziness, particularly avoidance of environments that provoke dizziness, dependence on the visual system, and excessive monitoring of bodily sensations. Patients develop alternative strategies for responding to symptoms of dizziness or unsteadiness, such as relaxation or distraction techniques. With systematic desensitization exposure response prevention (SDERP) treatment, gradual exposure to provocative environments is essential, enabling patients to habituate to, rather than avoid, symptoms.

Biofeedback (BFB) therapy is a noninvasive intervention through which individuals receive information on their physiological responses and learn to modify them actively. For example, Heart rate variability (HRV) BFB has recently been shown to be an effective intervention for a variety of psychophysiological disorders. The goal of BFB is for patients to gain a strong understanding of their physiological responses to environments around them and leverage that knowledge to lessen the severity and frequency of symptoms.

Given the vital role that visual inputs play in developing and perpetuating chronic dizziness, habituation to visual stimuli must be a significant component of treatment. However, visually provoked symptoms, rather than motion or position-provoked symptoms, are often the most resistant to current treatment options. One cause may be that visual stimuli are difficult to replicate in the clinic or office. As a result, using SDERP with a fear of symptom hierarchy in these visually stimulating environments cannot be fully addressed in these controlled treatment settings. One way to address this treatment gap is through virtual reality (VR) technology. VR immerses patients in realistic visual environments, making the exposure (in vivo) in real time a valuable adjunct to treatment.

Although VR has not been explicitly described in the treatment of PPPD, it has been piloted in the rehabilitation of peripheral vestibular dysfunction. These studies often employed large virtual reality theaters with multiple projected screens, and participants performed exercises while immersed in the environment. Preliminary studies have shown these VR interventions to be effective, particularly in reducing the severity of visually induced symptoms. Therefore, the current study hypothesizes that integrating VR into current PPPD treatment techniques - specifically BFB, SDERP, and CBT - may benefit patients and further strengthen the effectiveness of these methodologies. We will use a commercially available VR headset, which will enable the use of VR in the office setting and is a relatively low-cost form of VR technology. This study aims to evaluate the feasibility and effectiveness of VR in conjunction with BFB, SDERP, and CBT to investigate if VR technology will enhance the known effective treatments to reduce dizziness as a treatment approach to PPPD and other forms of chronic dizziness.

ELIGIBILITY:
Inclusion Criteria:

- Patients who previously or are currently seen in our program who have not already undergone BFB, CBT, and SDERP for treatment of their chronic dizziness.

Exclusion Criteria:

* Patients without chronic dizziness.
* Patients for whom written consent is not available.
* Patients who exhibit psychotic features, have untreated mental health conditions, or have an intellectual disability, developmental delay, or decisional impairment.
* Non-English language preference patients.
* Patients with a history of seizures, at risk of seizures, or who have a diagnosis of epilepsy.

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Dizziness Handicap Inventory | 1 year
  A 25-item self-assessment that quantifies the impact of dizziness on daily functioning. The DHI measures self-perceived handicap due to dizziness in the functional, emotional, and physical domains. Higher score corresponds to a greater perceived handicap due to dizziness.
Nijmegen Questionnaire | 1 year
  A 16-item self-report questionnaire to assess hyperventilation syndrome. Participants are asked to rate the occurrence of 16 symptoms commonly associated with hyperventilation syndrome on a 5-point Likert scale (0-Never; 4-Very often). A score greater than 23 suggests positive diagnosis of hyperventilation syndrome.
Pediatric Quality of Life Inventory | 1 year
  A 23-item inventory that measures health-related quality of life. The PedsQL consists of 4 scales: physical, emotional, social, school. Participants rate how often each item has been a problem for them within the past month on a 5-point Likert scale (0-Never; 4-Almost always). Higher score suggests lower health-related quality of life.
Fear of Pain Questionnaire | 1 year
  A 23 or 24-item (depending on self-report or parent-proxy version) questionnaire that assesses pain-related fears. Participants are asked to rate each item on a 5-point Likert scale (0-Strongly Disagree; 4-Strongly Agree). Higher score suggests a higher level of pain-related fears.
PROMIS Anxiety Measure | 1 year
  An 8-item self-report measure that screens for an quantifies the severity of anxiety symptoms. Participants rate the frequency of each item within the past seven days on a 5-point Likert scale (1-Never; 5-Almost always). A higher score suggests a higher severity of anxiety.
PROMIS Depression Measure | 1 year
  An 8-item self-report measure that screens for and quantifies the severity of depression symptoms. Participants rate the frequency of each item within the past seven days on a 5-point Likert scale (1-Never; 5-Always). Higher score suggests a higher severity of depression.
Niigata PPPD Questionnaire | 1 year
  A 12-item self-reported measure intended to assess symptom severity, specifically for PPPD. Participants rate how much eat item has affected them in the past week on a 7-point Likert scale (0-None; 6-Unbearable).

SECONDARY OUTCOMES:
Ratings of dizziness and pain severity, duration, and frequency | 1 year
  Each patient will have a "Chronic Dizziness Log" that subjectively tracks self-reported dizziness and pain associated with PPPD, including severity, duration, and frequency. Participants will be asked to report each measure on a scale of 1-10. (1-Not present; 10-As bad as it can be).
Degree of stress before, during, and after exposure to virtual environments | 1 year
  When experiencing a virtual reality (VR) environment via the VR headset, participants will be asked to report their level of stress before entering the environment, while in the environment, and after the exposure is over. Participants will be asked to report their stress on a scale of 1-10 (1-Not present; 10-As bad as it can be).
Degree of symptoms before, during, and after exposure to virtual environments | 1 year
  Each participant will be asked to report both the duration and the severity of their symptoms before entering a virtual reality environment, while experiencing that environment, and after the virtual reality exposure is over. They will be asked to report these symptom measures on a scale of 1-10 (1-Not present; 10-As bad as it can be).
Heart Rate Variability | 1 year
  A core component of biofeedback (BFB) therapy, HRV is the variation in time between each cardiac cycle, measured by ECG leads placed on the wrists and hands. This BFB measure allows researchers to track participants' progress in BFB therapy over time. HRV is expected to increase with successful treatment.
Respiratory Rate | 1 year
  A component of biofeedback (BFB) therapy, respiratory rate is the number of breaths per minute, measured by a flexible band that wraps around the participant's torso. Respiratory rate allows researchers to track participants' progress in BFB therapy.
Electrodermal Activity (Skin Conductance) | 1 year
  A component of biofeedback (BFB) therapy, electrodermal activity is the electrical conductivity of the skin, measured by small electrodes placed on the participant's fingers. Electrodermal activity allows researchers to measure the participants' progress in BFB therapy and relative level of stress/arousal.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob R Brodsky, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital at Waltham, Waltham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oh H, Lee G. Feasibility of full immersive virtual reality video game on balance and cybersickness of healthy adolescents. Neurosci Lett. 2021 Aug 24;760:136063. doi: 10.1016/j.neulet.2021.136063. Epub 2021 Jun 24. PMID 34174345
- [Background] Kim H, Kim DJ, Chung WH, Park KA, Kim JDK, Kim D, Kim K, Jeon HJ. Clinical predictors of cybersickness in virtual reality (VR) among highly stressed people. Sci Rep. 2021 Jun 9;11(1):12139. doi: 10.1038/s41598-021-91573-w. PMID 34108520
- [Background] Walker LS, Greene JW. The functional disability inventory: measuring a neglected dimension of child health status. J Pediatr Psychol. 1991 Feb;16(1):39-58. doi: 10.1093/jpepsy/16.1.39. PMID 1826329
- [Background] Yagi C, Morita Y, Kitazawa M, Nonomura Y, Yamagishi T, Ohshima S, Izumi S, Takahashi K, Horii A. A Validated Questionnaire to Assess the Severity of Persistent Postural-Perceptual Dizziness (PPPD): The Niigata PPPD Questionnaire (NPQ). Otol Neurotol. 2019 Aug;40(7):e747-e752. doi: 10.1097/MAO.0000000000002325. PMID 31219964
- [Background] Schalet BD, Pilkonis PA, Yu L, Dodds N, Johnston KL, Yount S, Riley W, Cella D. Clinical validity of PROMIS Depression, Anxiety, and Anger across diverse clinical samples. J Clin Epidemiol. 2016 May;73:119-27. doi: 10.1016/j.jclinepi.2015.08.036. Epub 2016 Feb 27. PMID 26931289
- [Background] Simons LE, Sieberg CB, Carpino E, Logan D, Berde C. The Fear of Pain Questionnaire (FOPQ): assessment of pain-related fear among children and adolescents with chronic pain. J Pain. 2011 Jun;12(6):677-86. doi: 10.1016/j.jpain.2010.12.008. Epub 2011 Feb 26. PMID 21354866
- [Background] Varni JW, Seid M, Rode CA. The PedsQL: measurement model for the pediatric quality of life inventory. Med Care. 1999 Feb;37(2):126-39. doi: 10.1097/00005650-199902000-00003. PMID 10024117
- [Background] van Dixhoorn J, Duivenvoorden HJ. Efficacy of Nijmegen Questionnaire in recognition of the hyperventilation syndrome. J Psychosom Res. 1985;29(2):199-206. doi: 10.1016/0022-3999(85)90042-x. PMID 4009520
- [Background] Jacobson GP, Newman CW. The development of the Dizziness Handicap Inventory. Arch Otolaryngol Head Neck Surg. 1990 Apr;116(4):424-7. doi: 10.1001/archotol.1990.01870040046011. PMID 2317323
- [Background] Pavlou M, Kanegaonkar RG, Swapp D, Bamiou DE, Slater M, Luxon LM. The effect of virtual reality on visual vertigo symptoms in patients with peripheral vestibular dysfunction: a pilot study. J Vestib Res. 2012;22(5-6):273-81. doi: 10.3233/VES-120462. PMID 23302708
- [Background] Alahmari KA, Sparto PJ, Marchetti GF, Redfern MS, Furman JM, Whitney SL. Comparison of virtual reality based therapy with customized vestibular physical therapy for the treatment of vestibular disorders. IEEE Trans Neural Syst Rehabil Eng. 2014 Mar;22(2):389-99. doi: 10.1109/TNSRE.2013.2294904. PMID 24608691
- [Background] Nolan RP, Liu S, Shoemaker JK, Hachinski V, Lynn H, Mikulis DJ, Wennberg RA, Moy Lum-Kwong M, Zbib A. Therapeutic benefit of internet-based lifestyle counselling for hypertension. Can J Cardiol. 2012 May;28(3):390-6. doi: 10.1016/j.cjca.2012.02.012. Epub 2012 Apr 11. PMID 22498181
- [Background] Nolan RP, Floras JS, Harvey PJ, Kamath MV, Picton PE, Chessex C, Hiscock N, Powell J, Catt M, Hendrickx H, Talbot D, Chen MH. Behavioral neurocardiac training in hypertension: a randomized, controlled trial. Hypertension. 2010 Apr;55(4):1033-9. doi: 10.1161/HYPERTENSIONAHA.109.146233. Epub 2010 Mar 1. PMID 20194302
- [Background] McCraty R, Atkinson M, Tomasino D. Impact of a workplace stress reduction program on blood pressure and emotional health in hypertensive employees. J Altern Complement Med. 2003 Jun;9(3):355-69. doi: 10.1089/107555303765551589. PMID 12816624
- [Background] Joseph CN, Porta C, Casucci G, Casiraghi N, Maffeis M, Rossi M, Bernardi L. Slow breathing improves arterial baroreflex sensitivity and decreases blood pressure in essential hypertension. Hypertension. 2005 Oct;46(4):714-8. doi: 10.1161/01.HYP.0000179581.68566.7d. Epub 2005 Aug 29. PMID 16129818
- [Background] Hallman DM, Olsson EM, von Scheele B, Melin L, Lyskov E. Effects of heart rate variability biofeedback in subjects with stress-related chronic neck pain: a pilot study. Appl Psychophysiol Biofeedback. 2011 Jun;36(2):71-80. doi: 10.1007/s10484-011-9147-0. PMID 21365308
- [Background] Siepmann M, Aykac V, Unterdorfer J, Petrowski K, Mueck-Weymann M. A pilot study on the effects of heart rate variability biofeedback in patients with depression and in healthy subjects. Appl Psychophysiol Biofeedback. 2008 Dec;33(4):195-201. doi: 10.1007/s10484-008-9064-z. Epub 2008 Sep 19. PMID 18807175
- [Background] Karavidas MK, Lehrer PM, Vaschillo E, Vaschillo B, Marin H, Buyske S, Malinovsky I, Radvanski D, Hassett A. Preliminary results of an open label study of heart rate variability biofeedback for the treatment of major depression. Appl Psychophysiol Biofeedback. 2007 Mar;32(1):19-30. doi: 10.1007/s10484-006-9029-z. Epub 2007 Mar 1. PMID 17333315
- [Background] Henriques G, Keffer S, Abrahamson C, Horst SJ. Exploring the effectiveness of a computer-based heart rate variability biofeedback program in reducing anxiety in college students. Appl Psychophysiol Biofeedback. 2011 Jun;36(2):101-12. doi: 10.1007/s10484-011-9151-4. PMID 21533678
- [Background] Riccelli R, Passamonti L, Toschi N, Nigro S, Chiarella G, Petrolo C, Lacquaniti F, Staab JP, Indovina I. Altered Insular and Occipital Responses to Simulated Vertical Self-Motion in Patients with Persistent Postural-Perceptual Dizziness. Front Neurol. 2017 Oct 17;8:529. doi: 10.3389/fneur.2017.00529. eCollection 2017. PMID 29089920
- [Background] Staab JP. Persistent Postural-Perceptual Dizziness. Semin Neurol. 2020 Feb;40(1):130-137. doi: 10.1055/s-0039-3402736. Epub 2020 Jan 14. PMID 31935771
- [Background] Huppert D, Strupp M, Rettinger N, Hecht J, Brandt T. Phobic postural vertigo--a long-term follow-up (5 to 15 years) of 106 patients. J Neurol. 2005 May;252(5):564-9. doi: 10.1007/s00415-005-0699-x. Epub 2005 Mar 4. PMID 15742115
- [Background] Wang A, Fleischman KM, Kawai K, Corcoran M, Brodsky JR. Persistent Postural-Perceptual Dizziness in Children and Adolescents. Otol Neurotol. 2021 Sep 1;42(8):e1093-e1100. doi: 10.1097/MAO.0000000000003212. PMID 34191779
- [Background] Wang A, Zhou G, Lipson S, Kawai K, Corcoran M, Brodsky JR. Multifactorial Characteristics of Pediatric Dizziness and Imbalance. Laryngoscope. 2021 Apr;131(4):E1308-E1314. doi: 10.1002/lary.29024. Epub 2020 Aug 18. PMID 32809223
- [Background] Staab JP, Ruckenstein MJ. Expanding the differential diagnosis of chronic dizziness. Arch Otolaryngol Head Neck Surg. 2007 Feb;133(2):170-6. doi: 10.1001/archotol.133.2.170. PMID 17309987
- [Background] Richmond RC, Tepper CS. Genetic and hormonal regulation of esterase 6 activity in male Drosophila melanogaster. Isozymes Curr Top Biol Med Res. 1983;9:91-106. PMID 6413454
- See also: Related Info — https://icd.who.int/browse/2025-01/mms/en